CLINICAL TRIAL: NCT05583058
Title: Sex Hormone Overdose and Misuse in Chinese Transgender and Gender Non-conforming Population: a Mixed-methods Study
Brief Title: Sex Hormone Overdose and Misuse in Chinese Transgender and Gender Non-conforming Population
Acronym: HODMChina
Status: Not yet recruiting | Type: Observational
Sponsor: Xiamen University (Other)
Collaborators: Tongji University (Other); Tsinghua University (Other)
Responsible Party: Principal Investigator, Ben-tuo Zeng, Principal Investigator, Xiamen University
Other Study IDs: HODM-TGNC-C-01O
Record Dates: First submitted 2022-10-10; First posted 2022-10-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Gender Incongruence; Gender Dysphoria
Keywords: Transgender Persons; Gender Affirming Hormone Therapy; Gender Dysphoria; Drug Overdose
MeSH Terms: conditions — Gender Dysphoria; Drug Overdose

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hormone Overdose and Misuse Group: Transgender and gender non-conforming individuals who have been identified as hormone overdose and misuse (HODM) at start of the cohorts according to the criteria established by the study.
  Interventions: Other: Hormone Overdose and Misuse
- Non-Hormone Overdose and Misuse Group: Transgender and gender non-conforming individuals who have been identified as without hormone overdose or misuse (HODM) at start of the cohorts according to the criteria established by the study.

INTERVENTIONS:
Other: Hormone Overdose and Misuse — This is an observational study. Hormone Overdose and Misuse is an exposure.
  Groups: Hormone Overdose and Misuse Group

SUMMARY:
The investigators propose to investigate the definition of hormone overdose and misuse (HODM) in Chinese transgender and gender nonconforming population (TGNCs), address the incidence of HODM in Chinese TGNC population, related factors and risks, identify the probable causes of HODM, and follow up HODM individuals to explore long-term effects.

The research questions are:

Q1 What is the definition and the criteria of HODM in Chinese TGNC population? Q2 What is the prevalence of HODM in Chinese TGNC population? Q3 What factors and risks are relevant to HODM? Q4 What are the causes? Q5 What are the long-term effects of HODM in Chinese TGNC population, compared to those who enroll in regular GAHT regimens?

The investigators decide to employ a mixed-methods design to construct a full research framework on HODM. A prospective cohort study is a component of the study.

The study can be divided into four stages to address research questions. Stage I will establish a precise definition and eligibility criteria of HODM through expert panel meeting and stakeholder engagement. Subsequently, a cross-sectional study will be conducted to evaluate the rate, subtypes, and related factors of HODM in Chinese TGNCs. In Stage III, semi-structured interviews and focus groups for TGNCs who are identified as HODM will be employed to investigate the causes, motivations and personal impact factors. This stage will be divided into two phases, Stage III-a before the cross-sectional study to provide a brief picture of HODM behaviors, and Stage III-b after the cross-sectional study to draw an overall pattern. Lastly, all participants of Stage II or III who would like to participate in our follow-up will be included in prospective cohorts to assess long-term effects.

Among the stages, the cohort study is the subject of the registration. The investigators propose two cohorts in the study. Participants who are identified as HODM will be assigned to cohort 1 [HODM cohort], and those who are identified as regular GAHT use will be assigned to cohort 2 [non-HODM cohort]. Participants will be asked to report their gender-related and hormone use-related conditions, and mental health-related conditions at specific timepoints. The investigators will compare the HODM cohort to the non-HODM cohort to see if the overall incidence of adverse effects, gender-related, hormone-related, and mental health-related conditions differ in the cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with Chinese nationality (excluding Hong Kong SAR, Macau SAR, and Taiwan).
* Aged over 12.
* Identify themselves as TGNCs of any subtypes, including transgender female, transgender male, genderqueer, gender non-binary, crossdresser, or other subtypes.
* have experienced at least one month of GAHT of any regimens and frequency in the last one year, or is taking hormones during the period of the study.
* Hormones taken include androgen, estrogen, progesterone, anti-androgen, and anti-estrogen of any chemical structures, trade names, or regimens.

Exclusion Criteria:

* Individuals who undertake GAHT in the absence of self-consciousness due to mental disorders, or under external coercion/abuse.
* Refuse to sign or unable to understand the informed consent.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Only individuals who identified themselves as transgender female, transgender male, genderqueer, gender non-binary, crossdresser, or any other subgroups of Transgender and Gender Non-conforming population (TGNCs) will be recruited.
Study Population: We will disseminate a questionnaire among online TGNC communities, social medias, under the help of TGNC-related non-government organizations (NGO). Each participant will be asked to share the link to other TGNCs. Only the completers of the questionnaire who agree to be followed up will be eligible for the cohort study. However, if needed, we will also recruit more TGNCs from outside previous participants via social media.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2022-12-15 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Moderate-to-severe adverse events | 24 months from the baseline assessment
  Any adverse events of Grade 2 or higher in Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. CTCAE v5.0 grades adverse effects as from grade 1 (asymptomatic or mild) to grade 5 (death).
Moderate-to-severe adverse events | 60 months from the baseline assessment
  Any adverse events of Grade 2 or higher in Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. CTCAE v5.0 grades adverse effects as from grade 1 (asymptomatic or mild) to grade 5 (death).

SECONDARY OUTCOMES:
GAHT attrition | 24 months from the baseline assessment
  Gender affirming hormone treatment attrition due to moderate-to-severe adverse events [any adverse events of Grade 2 or higher in Common Terminology Criteria for Adverse Events (CTCAE) version 5.0].
GAHT attrition | 60 months from the baseline assessment
  Gender affirming hormone treatment attrition due to moderate-to-severe adverse events [any adverse events of Grade 2 or higher in Common Terminology Criteria for Adverse Events (CTCAE) version 5.0].
Gender dysphoria | 24 months from the baseline assessment
  Gender dysphoria, evaluated using Utrecht Gender Dysphoria Scale - Gender Spectrum (UGDS-GS). UGDS-GS scores range from 18 to 90, and higher scores indicate higher levels of gender dysphoria.
Gender dysphoria | 60 months from the baseline assessment
  Gender dysphoria, evaluated using Utrecht Gender Dysphoria Scale - Gender Spectrum (UGDS-GS). UGDS-GS scores range from 18 to 90, and higher scores indicate higher levels of gender dysphoria.
Depression | 12 months from the baseline assessment
  Depression, evaluated using Patient Health Questionnaire-9 (PHQ-9) scale. PHQ-9 scores range from 0 to 27, and higher scores indicate higher levels of depression.
Depression | 24 months from the baseline assessment
  Depression, evaluated using Patient Health Questionnaire-9 (PHQ-9) scale. PHQ-9 scores range from 0 to 27, and higher scores indicate higher levels of depression.
Depression | 36 months from the baseline assessment
  Depression, evaluated using Patient Health Questionnaire-9 (PHQ-9) scale. PHQ-9 scores range from 0 to 27, and higher scores indicate higher levels of depression.
Depression | 60 months from the baseline assessment
  Depression, evaluated using Patient Health Questionnaire-9 (PHQ-9) scale. PHQ-9 scores range from 0 to 27, and higher scores indicate higher levels of depression.
Anxiety | 12 months from the baseline assessment
  Anxiety, evaluated using General Anxiety Disorder-7 (GAD-7) scale. GAD-7 scores range from 0 to 27, and higher scores indicate higher levels of anxiety.
Anxiety | 24 months from the baseline assessment
  Anxiety, evaluated using General Anxiety Disorder-7 (GAD-7) scale. GAD-7 scores range from 0 to 27, and higher scores indicate higher levels of anxiety.
Anxiety | 36 months from the baseline assessment
  Anxiety, evaluated using General Anxiety Disorder-7 (GAD-7) scale. GAD-7 scores range from 0 to 27, and higher scores indicate higher levels of anxiety.
Anxiety | 60 months from the baseline assessment
  Anxiety, evaluated using General Anxiety Disorder-7 (GAD-7) scale. GAD-7 scores range from 0 to 27, and higher scores indicate higher levels of anxiety.
General quality of life | 24 months from the baseline assessment
  Quality of life, using 36-Item Short Form Survey (SF-36) scale. SF-36 scores range from 0 to 100, and higher scores indicate better quality of life.
General quality of life | 60 months from the baseline assessment
  Quality of life, using 36-Item Short Form Survey (SF-36) scale. SF-36 scores range from 0 to 100, and higher scores indicate better quality of life.
Body image | 24 months from the baseline assessment
  Body image, using Body Image States Scale (BISS). BISS scores range from 6 to 54, and higher scores indicate worse body images.
Body image | 60 months from the baseline assessment
  Body image, using Body Image States Scale (BISS). BISS scores range from 6 to 54, and higher scores indicate worse body images.
Body-gender congruence | 24 months from the baseline assessment
  Body-gender congruence, evaluated using Transgender Congruence Scale (TCS). TCS scores range from 1 to 5 (or 12 to 60), and higher scores indicate better gender congruence.
Body-gender congruence | 60 months from the baseline assessment
  Body-gender congruence, evaluated using Transgender Congruence Scale (TCS). TCS scores range from 1 to 5 (or 12 to 60), and higher scores indicate better gender congruence.
Tanner stage | 12 months from the baseline assessment
  Tanner stages, evaluated using Visual Analogue Scale and Tanner Stage figures. Tanner stages divide the puberty process into 5 stages (stage 1 to stage 5), and higher stages indicate higher levels of puberty.
Tanner stage | 24 months from the baseline assessment
  Tanner stages, evaluated using Visual Analogue Scale and Tanner Stage figures. Tanner stages divide the puberty process into 5 stages (stage 1 to stage 5), and higher stages indicate higher levels of puberty.
Tanner stage | 36 months from the baseline assessment
  Tanner stages, evaluated using Visual Analogue Scale and Tanner Stage figures. Tanner stages divide the puberty process into 5 stages (stage 1 to stage 5), and higher stages indicate higher levels of puberty.
Gender identity | 24 months from the baseline assessment
  Gender identity, evaluated using Visual Analogue Scale, ranging from 0% female to 100% female. This score does not indicate any better or worse conditions.
Gender identity | 60 months from the baseline assessment
  Gender identity, evaluated using Visual Analogue Scale, ranging from 0% female to 100% female. This score does not indicate any better or worse conditions.

OTHER OUTCOMES:
Moderate-to-severe adverse events | 1 month from the baseline assessment
  Any adverse events of Grade 2 or higher in Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. CTCAE v5.0 grades adverse effects as from grade 1 (asymptomatic or mild) to grade 5 (death).
Moderate-to-severe adverse events | 3 months from the baseline assessment
  Any adverse events of Grade 2 or higher in Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. CTCAE v5.0 grades adverse effects as from grade 1 (asymptomatic or mild) to grade 5 (death).
Moderate-to-severe adverse events | 6 months from the baseline assessment
  Any adverse events of Grade 2 or higher in Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. CTCAE v5.0 grades adverse effects as from grade 1 (asymptomatic or mild) to grade 5 (death).
Moderate-to-severe adverse events | 12 months from the baseline assessment
  Any adverse events of Grade 2 or higher in Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. CTCAE v5.0 grades adverse effects as from grade 1 (asymptomatic or mild) to grade 5 (death).
Moderate-to-severe adverse events | 18 months from the baseline assessment
  Any adverse events of Grade 2 or higher in Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. CTCAE v5.0 grades adverse effects as from grade 1 (asymptomatic or mild) to grade 5 (death).
Moderate-to-severe adverse events | 30 months from the baseline assessment
  Any adverse events of Grade 2 or higher in Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. CTCAE v5.0 grades adverse effects as from grade 1 (asymptomatic or mild) to grade 5 (death).
Moderate-to-severe adverse events | 36 months from the baseline assessment
  Any adverse events of Grade 2 or higher in Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. CTCAE v5.0 grades adverse effects as from grade 1 (asymptomatic or mild) to grade 5 (death).
Moderate-to-severe adverse events | 42 months from the baseline assessment
  Any adverse events of Grade 2 or higher in Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. CTCAE v5.0 grades adverse effects as from grade 1 (asymptomatic or mild) to grade 5 (death).
Moderate-to-severe adverse events | 48 months from the baseline assessment
  Any adverse events of Grade 2 or higher in Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. CTCAE v5.0 grades adverse effects as from grade 1 (asymptomatic or mild) to grade 5 (death).
Moderate-to-severe adverse events | 54 months from the baseline assessment
  Any adverse events of Grade 2 or higher in Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. CTCAE v5.0 grades adverse effects as from grade 1 (asymptomatic or mild) to grade 5 (death).
GAHT attrition | 6 months from the baseline assessment
  Gender affirming hormone treatment attrition due to moderate-to-severe adverse events [any adverse events of Grade 2 or higher in Common Terminology Criteria for Adverse Events (CTCAE) version 5.0].
GAHT attrition | 12 months from the baseline assessment
  Gender affirming hormone treatment attrition due to moderate-to-severe adverse events [any adverse events of Grade 2 or higher in Common Terminology Criteria for Adverse Events (CTCAE) version 5.0].
GAHT attrition | 18 months from the baseline assessment
  Gender affirming hormone treatment attrition due to moderate-to-severe adverse events [any adverse events of Grade 2 or higher in Common Terminology Criteria for Adverse Events (CTCAE) version 5.0].
GAHT attrition | 30 months from the baseline assessment
  Gender affirming hormone treatment attrition due to moderate-to-severe adverse events [any adverse events of Grade 2 or higher in Common Terminology Criteria for Adverse Events (CTCAE) version 5.0].
GAHT attrition | 36 months from the baseline assessment
  Gender affirming hormone treatment attrition due to moderate-to-severe adverse events [any adverse events of Grade 2 or higher in Common Terminology Criteria for Adverse Events (CTCAE) version 5.0].
GAHT attrition | 42 months from the baseline assessment
  Gender affirming hormone treatment attrition due to moderate-to-severe adverse events [any adverse events of Grade 2 or higher in Common Terminology Criteria for Adverse Events (CTCAE) version 5.0].
GAHT attrition | 48 months from the baseline assessment
  Gender affirming hormone treatment attrition due to moderate-to-severe adverse events [any adverse events of Grade 2 or higher in Common Terminology Criteria for Adverse Events (CTCAE) version 5.0].
GAHT attrition | 54 months from the baseline assessment
  Gender affirming hormone treatment attrition due to moderate-to-severe adverse events [any adverse events of Grade 2 or higher in Common Terminology Criteria for Adverse Events (CTCAE) version 5.0].
Gender dysphoria | 3 months from the baseline assessment
  Gender dysphoria, evaluated using Utrecht Gender Dysphoria Scale - Gender Spectrum (UGDS-GS). UGDS-GS scores range from 18 to 90, and higher scores indicate higher levels of gender dysphoria.
Gender dysphoria | 6 months from the baseline assessment
  Gender dysphoria, evaluated using Utrecht Gender Dysphoria Scale - Gender Spectrum (UGDS-GS). UGDS-GS scores range from 18 to 90, and higher scores indicate higher levels of gender dysphoria.
Gender dysphoria | 12 months from the baseline assessment
  Gender dysphoria, evaluated using Utrecht Gender Dysphoria Scale - Gender Spectrum (UGDS-GS). UGDS-GS scores range from 18 to 90, and higher scores indicate higher levels of gender dysphoria.
Gender dysphoria | 18 months from the baseline assessment
  Gender dysphoria, evaluated using Utrecht Gender Dysphoria Scale - Gender Spectrum (UGDS-GS). UGDS-GS scores range from 18 to 90, and higher scores indicate higher levels of gender dysphoria.
Gender dysphoria | 30 months from the baseline assessment
  Gender dysphoria, evaluated using Utrecht Gender Dysphoria Scale - Gender Spectrum (UGDS-GS). UGDS-GS scores range from 18 to 90, and higher scores indicate higher levels of gender dysphoria.
Gender dysphoria | 36 months from the baseline assessment
  Gender dysphoria, evaluated using Utrecht Gender Dysphoria Scale - Gender Spectrum (UGDS-GS). UGDS-GS scores range from 18 to 90, and higher scores indicate higher levels of gender dysphoria.
Gender dysphoria | 42 months from the baseline assessment
  Gender dysphoria, evaluated using Utrecht Gender Dysphoria Scale - Gender Spectrum (UGDS-GS). UGDS-GS scores range from 18 to 90, and higher scores indicate higher levels of gender dysphoria.
Gender dysphoria | 48 months from the baseline assessment
  Gender dysphoria, evaluated using Utrecht Gender Dysphoria Scale - Gender Spectrum (UGDS-GS). UGDS-GS scores range from 18 to 90, and higher scores indicate higher levels of gender dysphoria.
Gender dysphoria | 54 months from the baseline assessment
  Gender dysphoria, evaluated using Utrecht Gender Dysphoria Scale - Gender Spectrum (UGDS-GS). UGDS-GS scores range from 18 to 90, and higher scores indicate higher levels of gender dysphoria.
Depression | 1 month from the baseline assessment
  Depression, evaluated using Patient Health Questionnaire-9 (PHQ-9) scale. PHQ-9 scores range from 0 to 27, and higher scores indicate higher levels of depression.
Depression | 3 months from the baseline assessment
  Depression, evaluated using Patient Health Questionnaire-9 (PHQ-9) scale. PHQ-9 scores range from 0 to 27, and higher scores indicate higher levels of depression.
Depression | 6 months from the baseline assessment
  Depression, evaluated using Patient Health Questionnaire-9 (PHQ-9) scale. PHQ-9 scores range from 0 to 27, and higher scores indicate higher levels of depression.
Depression | 18 months from the baseline assessment
  Depression, evaluated using Patient Health Questionnaire-9 (PHQ-9) scale. PHQ-9 scores range from 0 to 27, and higher scores indicate higher levels of depression.
Depression | 30 months from the baseline assessment
  Depression, evaluated using Patient Health Questionnaire-9 (PHQ-9) scale. PHQ-9 scores range from 0 to 27, and higher scores indicate higher levels of depression.
Depression | 42 months from the baseline assessment
  Depression, evaluated using Patient Health Questionnaire-9 (PHQ-9) scale. PHQ-9 scores range from 0 to 27, and higher scores indicate higher levels of depression.
Depression | 48 months from the baseline assessment
  Depression, evaluated using Patient Health Questionnaire-9 (PHQ-9) scale. PHQ-9 scores range from 0 to 27, and higher scores indicate higher levels of depression.
Depression | 54 months from the baseline assessment
  Depression, evaluated using Patient Health Questionnaire-9 (PHQ-9) scale. PHQ-9 scores range from 0 to 27, and higher scores indicate higher levels of depression.
Anxiety | 1 month from the baseline assessment
  Anxiety, evaluated using General Anxiety Disorder-7 (GAD-7) scale. GAD-7 scores range from 0 to 27, and higher scores indicate higher levels of anxiety.
Anxiety | 3 months from the baseline assessment
  Anxiety, evaluated using General Anxiety Disorder-7 (GAD-7) scale. GAD-7 scores range from 0 to 27, and higher scores indicate higher levels of anxiety.
Anxiety | 6 months from the baseline assessment
  Anxiety, evaluated using General Anxiety Disorder-7 (GAD-7) scale. GAD-7 scores range from 0 to 27, and higher scores indicate higher levels of anxiety.
Anxiety | 18 months from the baseline assessment
  Anxiety, evaluated using General Anxiety Disorder-7 (GAD-7) scale. GAD-7 scores range from 0 to 27, and higher scores indicate higher levels of anxiety.
Anxiety | 30 months from the baseline assessment
  Anxiety, evaluated using General Anxiety Disorder-7 (GAD-7) scale. GAD-7 scores range from 0 to 27, and higher scores indicate higher levels of anxiety.
Anxiety | 42 months from the baseline assessment
  Anxiety, evaluated using General Anxiety Disorder-7 (GAD-7) scale. GAD-7 scores range from 0 to 27, and higher scores indicate higher levels of anxiety.
Anxiety | 48 months from the baseline assessment
  Anxiety, evaluated using General Anxiety Disorder-7 (GAD-7) scale. GAD-7 scores range from 0 to 27, and higher scores indicate higher levels of anxiety.
Anxiety | 54 months from the baseline assessment
  Anxiety, evaluated using General Anxiety Disorder-7 (GAD-7) scale. GAD-7 scores range from 0 to 27, and higher scores indicate higher levels of anxiety.
General quality of life | 6 months from the baseline assessment
  Quality of life, using 36-Item Short Form Survey (SF-36) scale. SF-36 scores range from 0 to 100, and higher scores indicate better quality of life.
General quality of life | 12 months from the baseline assessment
  Quality of life, using 36-Item Short Form Survey (SF-36) scale. SF-36 scores range from 0 to 100, and higher scores indicate better quality of life.
General quality of life | 18 months from the baseline assessment
  Quality of life, using 36-Item Short Form Survey (SF-36) scale. SF-36 scores range from 0 to 100, and higher scores indicate better quality of life.
General quality of life | 30 months from the baseline assessment
  Quality of life, using 36-Item Short Form Survey (SF-36) scale. SF-36 scores range from 0 to 100, and higher scores indicate better quality of life.
General quality of life | 36 months from the baseline assessment
  Quality of life, using 36-Item Short Form Survey (SF-36) scale. SF-36 scores range from 0 to 100, and higher scores indicate better quality of life.
General quality of life | 42 months from the baseline assessment
  Quality of life, using 36-Item Short Form Survey (SF-36) scale. SF-36 scores range from 0 to 100, and higher scores indicate better quality of life.
General quality of life | 48 months from the baseline assessment
  Quality of life, using 36-Item Short Form Survey (SF-36) scale. SF-36 scores range from 0 to 100, and higher scores indicate better quality of life.
General quality of life | 54 months from the baseline assessment
  Quality of life, using 36-Item Short Form Survey (SF-36) scale. SF-36 scores range from 0 to 100, and higher scores indicate better quality of life.
Body image | 6 months from the baseline assessment
  Body image, using Body Image States Scale (BISS). BISS scores range from 6 to 54, and higher scores indicate worse body images.
Body image | 12 months from the baseline assessment
  Body image, using Body Image States Scale (BISS). BISS scores range from 6 to 54, and higher scores indicate worse body images.
Body image | 18 months from the baseline assessment
  Body image, using Body Image States Scale (BISS). BISS scores range from 6 to 54, and higher scores indicate worse body images.
Body image | 30 months from the baseline assessment
  Body image, using Body Image States Scale (BISS). BISS scores range from 6 to 54, and higher scores indicate worse body images.
Body image | 36 months from the baseline assessment
  Body image, using Body Image States Scale (BISS). BISS scores range from 6 to 54, and higher scores indicate worse body images.
Body image | 42 months from the baseline assessment
  Body image, using Body Image States Scale (BISS). BISS scores range from 6 to 54, and higher scores indicate worse body images.
Body image | 48 months from the baseline assessment
  Body image, using Body Image States Scale (BISS). BISS scores range from 6 to 54, and higher scores indicate worse body images.
Body image | 54 months from the baseline assessment
  Body image, using Body Image States Scale (BISS). BISS scores range from 6 to 54, and higher scores indicate worse body images.
Body-gender congruence | 3 months from the baseline assessment
  Body-gender congruence, evaluated using Transgender Congruence Scale (TCS). TCS scores range from 1 to 5 (or 12 to 60), and higher scores indicate better gender congruence.
Body-gender congruence | 6 months from the baseline assessment
  Body-gender congruence, evaluated using Transgender Congruence Scale (TCS). TCS scores range from 1 to 5 (or 12 to 60), and higher scores indicate better gender congruence.
Body-gender congruence | 12 months from the baseline assessment
  Body-gender congruence, evaluated using Transgender Congruence Scale (TCS). TCS scores range from 1 to 5 (or 12 to 60), and higher scores indicate better gender congruence.
Body-gender congruence | 18 months from the baseline assessment
  Body-gender congruence, evaluated using Transgender Congruence Scale (TCS). TCS scores range from 1 to 5 (or 12 to 60), and higher scores indicate better gender congruence.
Body-gender congruence | 30 months from the baseline assessment
  Body-gender congruence, evaluated using Transgender Congruence Scale (TCS). TCS scores range from 1 to 5 (or 12 to 60), and higher scores indicate better gender congruence.
Body-gender congruence | 36 months from the baseline assessment
  Body-gender congruence, evaluated using Transgender Congruence Scale (TCS). TCS scores range from 1 to 5 (or 12 to 60), and higher scores indicate better gender congruence.
Body-gender congruence | 42 months from the baseline assessment
  Body-gender congruence, evaluated using Transgender Congruence Scale (TCS). TCS scores range from 1 to 5 (or 12 to 60), and higher scores indicate better gender congruence.
Body-gender congruence | 48 months from the baseline assessment
  Body-gender congruence, evaluated using Transgender Congruence Scale (TCS). TCS scores range from 1 to 5 (or 12 to 60), and higher scores indicate better gender congruence.
Body-gender congruence | 54 months from the baseline assessment
  Body-gender congruence, evaluated using Transgender Congruence Scale (TCS). TCS scores range from 1 to 5 (or 12 to 60), and higher scores indicate better gender congruence.
Tanner stage | 3 months from the baseline assessment
  Tanner stages, evaluated using Visual Analogue Scale and Tanner Stage figures. Tanner stages divide the puberty process into 5 stages (stage 1 to stage 5), and higher stages indicate higher levels of puberty.
Tanner stage | 6 months from the baseline assessment
  Tanner stages, evaluated using Visual Analogue Scale and Tanner Stage figures. Tanner stages divide the puberty process into 5 stages (stage 1 to stage 5), and higher stages indicate higher levels of puberty.
Tanner stage | 18 months from the baseline assessment
  Tanner stages, evaluated using Visual Analogue Scale and Tanner Stage figures. Tanner stages divide the puberty process into 5 stages (stage 1 to stage 5), and higher stages indicate higher levels of puberty.
Tanner stage | 30 months from the baseline assessment
  Tanner stages, evaluated using Visual Analogue Scale and Tanner Stage figures. Tanner stages divide the puberty process into 5 stages (stage 1 to stage 5), and higher stages indicate higher levels of puberty.
Tanner stage | 42 months from the baseline assessment
  Tanner stages, evaluated using Visual Analogue Scale and Tanner Stage figures. Tanner stages divide the puberty process into 5 stages (stage 1 to stage 5), and higher stages indicate higher levels of puberty.
Tanner stage | 48 months from the baseline assessment
  Tanner stages, evaluated using Visual Analogue Scale and Tanner Stage figures. Tanner stages divide the puberty process into 5 stages (stage 1 to stage 5), and higher stages indicate higher levels of puberty.
Tanner stage | 54 months from the baseline assessment
  Tanner stages, evaluated using Visual Analogue Scale and Tanner Stage figures. Tanner stages divide the puberty process into 5 stages (stage 1 to stage 5), and higher stages indicate higher levels of puberty.
Tanner stage | 60 months from the baseline assessment
  Tanner stages, evaluated using Visual Analogue Scale and Tanner Stage figures. Tanner stages divide the puberty process into 5 stages (stage 1 to stage 5), and higher stages indicate higher levels of puberty.
Gender identity | 3 months from the baseline assessment
  Gender identity, evaluated using Visual Analogue Scale, ranging from 0% female to 100% female. This score does not indicate any better or worse conditions.
Gender identity | 6 months from the baseline assessment
  Gender identity, evaluated using Visual Analogue Scale, ranging from 0% female to 100% female. This score does not indicate any better or worse conditions.
Gender identity | 12 months from the baseline assessment
  Gender identity, evaluated using Visual Analogue Scale, ranging from 0% female to 100% female. This score does not indicate any better or worse conditions.
Gender identity | 18 months from the baseline assessment
  Gender identity, evaluated using Visual Analogue Scale, ranging from 0% female to 100% female. This score does not indicate any better or worse conditions.
Gender identity | 30 months from the baseline assessment
  Gender identity, evaluated using Visual Analogue Scale, ranging from 0% female to 100% female. This score does not indicate any better or worse conditions.
Gender identity | 36 months from the baseline assessment
  Gender identity, evaluated using Visual Analogue Scale, ranging from 0% female to 100% female. This score does not indicate any better or worse conditions.
Gender identity | 42 months from the baseline assessment
  Gender identity, evaluated using Visual Analogue Scale, ranging from 0% female to 100% female. This score does not indicate any better or worse conditions.
Gender identity | 48 months from the baseline assessment
  Gender identity, evaluated using Visual Analogue Scale, ranging from 0% female to 100% female. This score does not indicate any better or worse conditions.
Gender identity | 54 months from the baseline assessment
  Gender identity, evaluated using Visual Analogue Scale, ranging from 0% female to 100% female. This score does not indicate any better or worse conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Ben-tuo Zeng, Principal Investigator — School of Medicine, Xiamen University
Locations (1):
- School of Medicine, Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study protocol — https://doi.org/10.1101/2022.10.05.22280725